CLINICAL TRIAL: NCT01868139
Title: A Phase II, Multi-Center Study of Interventional Spray Cryotherapy for Early-Stage Esophageal Cancer (ICE-CANCER)
Brief Title: Spray Cryotherapy for Esophageal Cancer (ICE-CANCER)
Acronym: ICE-CANCER
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: insufficient accrual
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Bruce Greenwald, Professor of Medicine, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HP-00052885
Record Dates: First submitted 2013-03-30; First posted 2013-06-04 (Estimated); Results first posted 2019-10-17 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2022-03

CONDITIONS: Esophageal Cancer
Keywords: Cryotherapy; Esophageal cancer; Esophageal carcinoma; Liquid nitrogen; Esophageal adenocarcinoma; Esophageal squamous cell carcinoma; Endoscopy; Ablation
MeSH Terms: conditions — Esophageal Neoplasms; Adenocarcinoma Of Esophagus; Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cryotherapy (Experimental): Liquid nitrogen spray cryotherapy with the truFreeze device
  Interventions: Device: Liquid nitrogen spray cryotherapy with the truFreeze device

INTERVENTIONS:
Device: Liquid nitrogen spray cryotherapy with the truFreeze device — Low-pressure liquid nitrogen is sprayed through an upper endoscope on the diseased esophageal tissue to freeze and destroy it. The upper endoscope enables direct visualization of mucosal freeze during spray of the liquid nitrogen onto the mucosa and avoids the need for direct contact with the tissues. The target area is frozen and thawed for several consecutive cycles. The treated tissue becomes necrotic and sloughs, with new, healthy tissue regenerating in its place.
  Other Names: truFreeze

SUMMARY:
The goal of this study is to evaluate the safety and efficacy of endoscopic spray cryotherapy using the CSA Medical, Inc. truFreeze System for patients with previously untreated early-stage cancer (T1a, N0, M0) who are ineligible or refuse conventional therapy including surgery, chemotherapy, radiation therapy, and endoscopic resection.

It is hypothesized that one of the two following outcomes will occur:

1. Complete response to therapy: complete tumor eradication confirmed through histologic examination of biopsy specimens from the targeted esophageal tissue site;
2. Stable disease: tumor remission is not attained, but disease progression is halted.

DETAILED DESCRIPTION:
Background

Endoscopic modalities have been reported to be effective in definitive treatment of early stage esophageal cancer. A study comparing endoscopic treatment to surgery in early esophageal cancer using the SEER (Surveillance Epidemiology and End Results) database showed no difference in the relative hazard of death from esophageal cancer between the two groups. The primary endoscopic therapies used in this study were endoscopic mucosal resection (EMR) and photodynamic therapy (PDT). Estimated 1 and 3 year survival in this study were 92% and 75% in the endoscopic arm and 92% and 82% in the surgical arm. EMR, endoscopic excision of superficial cancer, has also been shown to be highly effective in mucosal tumors in single center studies. "Low-risk" lesions, defined as flat or raised mucosal tumors 2 cm or less that are well-or moderately-differentiated without lymphovascular invasion, demonstrate complete response was seen in 96.6% of patients with 5 year survival of 84%. However, "high-risk lesions," defined as greater than 2 cm, poorly-differentiated, flat-ulcerated, or invading into the submucosa, have a complete remission rate of only 59%.

Endoscopic resection is not possible in all mucosal cancers. Some cancers are not visible endoscopically but detected only by endoscopic biopsy. In other cases, the EMR cannot be done due to scarring from previous resection or other therapy, especially external beam radiation. Management of these cases is problematic. PDT using porfimer sodium has been extensively studied for Barrett's esophagus with high-grade dysplasia, however studies of PDT for early stage esophageal cancer are limited. In a recent single site study using PDT and EMR for mucosal cancers, overall survival was comparable to a group treated with esophagectomy at the same center, with estimated 1 and 3 year survival of 98% and 95%. PDT was used in 43% in combination with EMR in the endoscopic treatment group. Recurrent carcinoma was detected in 16% of endoscopically treated patients. All recurrences were intramucosal cancers, with all but one managed by EMR. Overall, endoscopic treatment was well-tolerated. However, side effects of PDT are common and include photosensitivity, esophageal stricture, chest pain, nausea, vomiting, and fever. In the U.S., PDT is no longer commonly used in the esophagus due to availability of alternative treatment modalities with less cost and side effects.

Endoscopic spray cryotherapy with liquid nitrogen has emerged as an alternative treatment in stage I esophageal cancer in those not suitable for other therapies. A recent retrospective review at 10 U.S. centers assessed outcomes in seventy-nine patients. Patients included those with esophageal carcinoma who failed, refused, or were ineligible for conventional therapy including chemotherapy, radiation, combination chemotherapy and radiation, esophagectomy, and endoscopic mucosal resection. The majority of patients (76%) had tumor stage T1N0M0 with mean tumor length of 4 cm. All patients were treated with liquid nitrogen spray cryotherapy, and forty-nine patients completed treatment. Complete response of luminal disease occurred in 61.2%, including 18 of 24 (75%) with mucosal cancer. Follow-up averaged 10.6 to 11.5 months, and no serious adverse events were reported. Longer term follow-up was reported recently in abstract form. Complete response was seen in 92% of patients with mucosal cancer with median follow-up of 28 months and overall estimated survival at 1 and 3 years of 98% and 92% respectively.

Published studies have demonstrated spray cryotherapy to be safe and well-tolerated, with low overall complication rates. Tolerance of the procedure is very good. All procedures are performed on an outpatient basis. Primary side effects include chest pain, dysphagia, and odynophagia, reported in about half of all procedures. Mean duration of symptoms was 3.6 days, and many patients had no side effects after treatment. Serious adverse events were rare. Gastric perforation occurred in one patient with Marfan's syndrome. Benign esophageal stricture was reported in 13% of patients treated for cancer, with previous esophageal narrowing noted in 9/10. In combination with its relative cost-effectiveness and minimal invasiveness, endoscopic spray cryotherapy is an appealing option for those with stage I esophageal cancer who are ineligible or refuse conventional therapies.

Study Device: truFreezeTM System, CSA Medical Inc., Baltimore, MD

Study Objective: The objective of this study is to evaluate the safety and efficacy of endoscopic spray cryotherapy using the CSA Medical, Inc. truFreeze™ System for patients with early-stage esophageal cancer (T1a, N0, M0) who are ineligible or refuse conventional therapy including surgery, chemotherapy, radiation therapy, and endoscopic resection.

Study Design: Multi-center phase II study.

Study Population: Patients with early-stage esophageal cancer (stage T1aN0M0)

Study Duration: It is estimated that enrollment will take approximately two years. Each subject will remain in the study for up to one-year of treatment and for three years post-treatment. It is expected to take five years to collect all required data for this study.

Sample size: 40

Treatment

Participant receives liquid nitrogen spray cryotherapy every 4 - 8 weeks x no more than 8 cycles. Those with complete response to therapy will proceed to surveillance. Those with stable or responding disease will continue with cryotherapy. Those with progression of disease will discontinue protocol. For responding or stable disease after 8 cycles, continue treatment beyond 8 cycles until tumor progression or unacceptable toxicity. Discontinue protocol therapy for disease progression or unacceptable toxicity.

Follow-Up Evaluations and Data Collection

Patients will return for surveillance EGD (esophagogastroduodenoscopy) procedures with biopsies at 3, 6, 9, 12, 18, 24, 30, and 36 months (± 4 weeks) after the last cryotherapy treatment. An estimate of tumor size and response compared to baseline will be made at each endoscopy. Biopsies will be performed using large capacity forceps. In the area where tumor was present, biopsies will be taken every 1 cm in each quadrant. Directed biopsies will be performed in any areas that appear suspicious for cancer.

CT scan of the chest, abdomen, and pelvis (with oral and intravenous contrast if possible) will be performed every 6 months during the follow-up period. Full body PET/CT may also be performed instead of CT scanning.

Endoscopic ultrasound will be performed 6 months after treatment completion to assess for lymphadenopathy.

At the conclusion of this protocol, regardless of the outcome, patients will continue to require periodic surveillance endoscopies for re-emergence of esophageal cancer consistent with the standard surveillance guidelines. This monitoring will be performed at the investigator's site unless otherwise desired by the patient.

ELIGIBILITY:
Inclusion Criteria:

* T1aN0M0 esophageal cancer (tumor invades no deeper than lamina propria or muscularis mucosa, no regional lymph node or distant metastases), with the following minimum diagnostic workup:
* History/physical exam within 6 weeks prior to enrollment
* PET and CT scan of the chest and abdomen within 12 weeks prior to enrollment
* Endoscopy with histology or cytology confirming carcinoma
* Endoscopic ultrasound (EUS) with evaluation of the esophageal wall, mediastinum, and upper abdomen for evidence of abnormal lymph nodes. Suspicious lymph nodes will undergo EUS-guided fine needle aspiration if appropriate, as determined by the investigator.
* Endoscopic resection of focal lesions with histologic confirmation of positive deep margin or residual cancer within the esophagus
* Not a candidate for or refuses conventional therapies (surgery, radiation, chemotherapy, endoscopic resection) as determined by evaluation by the investigator, discussion with the patient, and review in Thoracic or Gastrointestinal Tumor Board.
* For females: not pregnant (negative pregnancy test within 14 days of starting study treatment), on acceptable means of contraception (oral contraceptives, barrier methods, approved contraceptive implant, long-term injectable contraception, intrauterine device or tubal ligation), or not of child bearing potential. Patients are considered not of child bearing potential if they are surgically sterile (they have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are postmenopausal.
* 18 years of age or older
* ECOG Performance Status 0 - 2

Exclusion Criteria:

* Medically unfit or other contraindication to tolerate upper endoscopy with ablation
* Contraindication to endoscopic spray cryotherapy as outlined in the directions for use for the device
* Other malignancy (except nonmelanoma skin cancer) within the past 1 year
* Co-morbid illness expected to cause death within 6 months
* Esophageal stricture preventing passage of endoscope or catheter
* Concurrent enrollment in an investigational drug or device trial that clinically interferes with this study's endpoints throughout the study
* Inability to provide informed consent or comply with this protocol
* Concurrent or previous cancer therapy for current esophageal malignancy by esophagectomy, chemotherapy, radiation therapy, and photodynamic therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2013-06; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce D Greenwald, MD, Principal Investigator — University of Maryland
Locations (1):
- University of Maryland Medical Center, Baltimore, Maryland, United States

REFERENCES:
- [Background] Greenwald BD, Dumot JA, Abrams JA, Lightdale CJ, David DS, Nishioka NS, Yachimski P, Johnston MH, Shaheen NJ, Zfass AM, Smith JO, Gill KR, Burdick JS, Mallat D, Wolfsen HC. Endoscopic spray cryotherapy for esophageal cancer: safety and efficacy. Gastrointest Endosc. 2010 Apr;71(4):686-93. doi: 10.1016/j.gie.2010.01.042. PMID 20363410
- [Background] Greenwald BD, et al. Spray cryotherapy for esophageal cancer: Long-term results. Am J Gastroenterol 2011;106:S7
- [Background] Greenwald BD, Dumot JA, Horwhat JD, Lightdale CJ, Abrams JA. Safety, tolerability, and efficacy of endoscopic low-pressure liquid nitrogen spray cryotherapy in the esophagus. Dis Esophagus. 2010 Jan;23(1):13-9. doi: 10.1111/j.1442-2050.2009.00991.x. Epub 2009 Jun 9. PMID 19515183
- [Background] Ribeiro A, et al. First report of spray cryosurgery depth of injury to the human esophagus. 2010. http://www.sages.org/meetings/annual_meeting/2010/resources/
- [Background] Gage AA, Baust J. Mechanisms of tissue injury in cryosurgery. Cryobiology. 1998 Nov;37(3):171-86. doi: 10.1006/cryo.1998.2115. PMID 9787063
- [Background] Johnston LR, Johnston MH. Cryo Spray Ablation (CSA) in the Esophagus: Optimization of Dosimetry. Am J Gastroenterol 2006;101:S532-533
- [Background] Das A, Singh V, Fleischer DE, Sharma VK. A comparison of endoscopic treatment and surgery in early esophageal cancer: an analysis of surveillance epidemiology and end results data. Am J Gastroenterol. 2008 Jun;103(6):1340-5. doi: 10.1111/j.1572-0241.2008.01889.x. Epub 2008 May 28. PMID 18510606
- [Background] Ell C, May A, Pech O, Gossner L, Guenter E, Behrens A, Nachbar L, Huijsmans J, Vieth M, Stolte M. Curative endoscopic resection of early esophageal adenocarcinomas (Barrett's cancer). Gastrointest Endosc. 2007 Jan;65(1):3-10. doi: 10.1016/j.gie.2006.04.033. PMID 17185072
- [Background] Ell C, May A, Gossner L, Pech O, Gunter E, Mayer G, Henrich R, Vieth M, Muller H, Seitz G, Stolte M. Endoscopic mucosal resection of early cancer and high-grade dysplasia in Barrett's esophagus. Gastroenterology. 2000 Apr;118(4):670-7. doi: 10.1016/s0016-5085(00)70136-3. PMID 10734018
- [Background] Overholt BF, Lightdale CJ, Wang KK, Canto MI, Burdick S, Haggitt RC, Bronner MP, Taylor SL, Grace MG, Depot M; International Photodynamic Group for High-Grade Dysplasia in Barrett's Esophagus. Photodynamic therapy with porfimer sodium for ablation of high-grade dysplasia in Barrett's esophagus: international, partially blinded, randomized phase III trial. Gastrointest Endosc. 2005 Oct;62(4):488-98. doi: 10.1016/j.gie.2005.06.047. PMID 16185958
- [Background] Overholt BF, Wang KK, Burdick JS, Lightdale CJ, Kimmey M, Nava HR, Sivak MV Jr, Nishioka N, Barr H, Marcon N, Pedrosa M, Bronner MP, Grace M, Depot M; International Photodynamic Group for High-Grade Dysplasia in Barrett's Esophagus. Five-year efficacy and safety of photodynamic therapy with Photofrin in Barrett's high-grade dysplasia. Gastrointest Endosc. 2007 Sep;66(3):460-8. doi: 10.1016/j.gie.2006.12.037. Epub 2007 Jul 23. PMID 17643436
- [Background] Pech O, Behrens A, May A, Nachbar L, Gossner L, Rabenstein T, Manner H, Guenter E, Huijsmans J, Vieth M, Stolte M, Ell C. Long-term results and risk factor analysis for recurrence after curative endoscopic therapy in 349 patients with high-grade intraepithelial neoplasia and mucosal adenocarcinoma in Barrett's oesophagus. Gut. 2008 Sep;57(9):1200-6. doi: 10.1136/gut.2007.142539. Epub 2008 May 6. PMID 18460553
- [Background] Prasad GA, Wu TT, Wigle DA, Buttar NS, Wongkeesong LM, Dunagan KT, Lutzke LS, Borkenhagen LS, Wang KK. Endoscopic and surgical treatment of mucosal (T1a) esophageal adenocarcinoma in Barrett's esophagus. Gastroenterology. 2009 Sep;137(3):815-23. doi: 10.1053/j.gastro.2009.05.059. Epub 2009 Jun 12. PMID 19524578

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment: Treated with liquid nitrogen spray cryotherapy
Period: Overall Study
Arm/Group | Treatment
Started | 1
Completed | 0
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Cryotherapy
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants] — Population: subject did not complete study
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Response Rate to Therapy
Description: The primary endpoint is to determine the response rate to spray cryotherapy.
  It is hypothesized that one of the two following outcomes will occur:
  1. Complete response to therapy: complete tumor eradication confirmed through histologic examination of biopsy specimens from the targeted esophageal tissue site;
  2. Stable disease: tumor remission is not attained, but disease progression is halted.
Time Frame: 5 years
Population: subject withdrawn before outcome measures could be assessed
Arm/Group | Treatment
Number analyzed (Participants) | 0

2. Secondary Outcome: Disease-free Survival at 12 Months After Treatment
Time Frame: 12 months
Population: subject withdrawn before outcome measures could be assessed
Arm/Group | Cryotherapy
Number analyzed (Participants) | 0

3. Secondary Outcome: Cancer Recurrence Rate at 12 Months After Treatment
Time Frame: 12 months
Population: subject withdrawn before outcome measures could be assessed
Arm/Group | Cryotherapy
Number analyzed (Participants) | 0

4. Secondary Outcome: Estimate Overall Survival
Time Frame: 12 months
Population: subject withdrawn before outcome measures could be assessed
Arm/Group | Cryotherapy
Number analyzed (Participants) | 0

5. Secondary Outcome: Estimate Progression-free Survival in Those Who do Not Achieve Complete Pathologic Response
Time Frame: 36 months
Population: subject withdrawn before outcome measures could be assessed
Arm/Group | Treatment
Number analyzed (Participants) | 0

6. Secondary Outcome: Number of Treatment Sessions Needed for Complete Response in Subjects in Whom the Primary Endpoint is Attained;
Time Frame: 12 months
Population: subject withdrawn before outcome measures could be assessed
Arm/Group | Treatment
Number analyzed (Participants) | 0

7. Secondary Outcome: Safety of Spray Cryotherapy in This Setting;
Description: Number of participants with adverse events; Number of adverse events within the study
Time Frame: 36 months
Population: subject withdrawn from study before outcomes measures could be assessed
Arm/Group | Treatment
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No